CLINICAL TRIAL: NCT05413798
Title: Clinical Performance Validation of Urine HPV Testing for Cervical Cancer Screening Among Women Living With HIV in South Africa
Brief Title: Urine HPV Testing for Cervical Cancer Screening Among Women Living With HIV in South Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IGHID12022; U54CA254564-01 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer; CIN2; CIN3
Keywords: cervical cancer; HPV; urine test; HIV
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Other): This is a single arm study. All participants will receive same interventions.
  Interventions: Other: Urine HPV testing; Other: Self-collected cervicovaginal specimen; Other: Provider-collected cervical samples

INTERVENTIONS:
Other: Urine HPV testing — Human papillomavirus (HPV) testing in urine sample.
Other: Self-collected cervicovaginal specimen — Human papillomavirus (HPV) testing in self-collected cervicovaginal specimen sample.
Other: Provider-collected cervical samples — Human papillomavirus (HPV) testing in healthcare provider collected cervicovaginal specimen sample.

SUMMARY:
The purpose of this study explores the usefulness of urine samples for cervical cancer screening in human immunodeficiency virus (HIV)-infected women.

Cervical cancer occurs when women are infected with the human papillomavirus (HPV), which can cause changes in the cells that lead to cervical precancer and, eventually, cervical cancer if untreated. However, urine HPV testing has not been well validated low- and middle-income country settings, with no data available to guide its use in HIV-infected women.

DETAILED DESCRIPTION:
Invasive cervical cancer is a significant health burden in low and middle income countries.

HIV-infected women in Africa are particularly affected and have an estimated invasive cervical cancer risk ~20-fold higher than women without HIV. Previous studies have been performed among only HIV-uninfected women or those whose HIV status was unknown. Additionally, HIV infected women are often diagnosed with invasive cervical cancer at younger ages.

Cervical cancer is preventable by regular screenings which includes doing a pap smear or HPV tests. There is also treatment of precancerous cervical lesions and vaccination against high risk types of HPV. World Health Organization currently recommends high risk HPV testing for cervical cancer screening in both high and low resources settings. National Guidelines in many low and middle income countries, including South Africa, have been updated to include plans to transition from cytology or visual screening to primary HPV screening. Urine HPV testing could provide a simpler approach for cervical screening that is more easily scaled in low and middle income countries.

The study hypothesizes that high-risk human papillomavirus (hrHPV) testing on urine specimens will be similar in sensitivity and specificity for the detection of cervical intra-epithelial neoplasia grade 2 or worse (CIN2+) compared to self- or clinician-collected sampling.

This study will investigate whether women can collect their own samples for HPV testing using either urine or a small brush in the vagina. The results of HPV tests on urine, self-collected vaginal samples, and provider-collected cervical samples will be compared to see which sample type works best.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. Confirmed HIV-1 infection
2. Age 25 years and older.
3. Be willing and able to provide written informed consent.

Exclusion Criteria:

1. Pregnant or intend to become pregnant within 90 days of enrollment
2. Have been screened for cervical cancer within the preceding year (365 days)
3. Have an active sexually transmitted infection (STI; women may participate once treated)
4. Have a surgically absent cervix
5. Have a history of cervical cancer
6. have been vaccinated against HPV.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is cervical cancer screening and targets only female participants.
Enrollment: 300 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of hrHPV testing in the three sample types for the detection of CIN2 | 4 weeks (Entry visit)
  The clinical performance (sensitivity, specificity, positive predictive value, and negative predictive value) for CIN2+ detection of sample collection methods namely urine, self-collected samples, and provider-collected samples will be determined.

SECONDARY OUTCOMES:
Clinical performance of hrHPV testing in in the three sample types for the detection of CIN3 or worse | 4 weeks
  The clinical performance (sensitivity, specificity, positive predictive value, and negative predictive value) for CIN3+ detection or worse of sample collection methods namely urine, self-collected samples, and provider-collected samples will be determined.
The proportion of participants positive for hrHPV | 4 weeks
  The high-risk human papillomavirus (hrHPV) positivity detection of urine, self-collected cervicovaginal specimen, and provider-collected cervical samples will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Chibwesha, MD, MSc, Principal Investigator — Division of Global Women's Health Department of Obstetrics and Gynecology, UNC Chapel Hill, NC
Locations (1):
- Clinical HIV Research Unit Temba Lethu Wing Helen Joseph Hospital, Westdene, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No
The rights and privacy of individuals who participate in research will be protected at all times. Thus, data intended for broader use will be stripped of identifiers that would permit linkages to individual research participants or variables that could lead to deductive disclosure of the identity of individual subjects. Research data that documents, supports and validates research findings will be made available after the main findings from the final research dataset have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers. All data sharing will abide by rules and/or policies defined by the sponsor, relevant IRBs, U.S. local, state, and federal laws and regulations, as well as South African laws and regulations.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials